CLINICAL TRIAL: NCT06684275
Title: Comparison of Pulsed and Thermal Radiofrequency for the Treatment of Trigeminal Neuralgia: A Randomized Controlled Trial
Brief Title: Comparison of Pulsed and Thermal Radiofrequency for Trigeminal Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Awad Bessar, Assistant Professor of Diagnostic and Interventional Radiology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRF-TRF-TN
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; Pulsed Radiofrequency; Thermal Radiofrequency; Neuropathic Pain; Facial Pain; Radiofrequency Ablation
MeSH Terms: conditions — Trigeminal Neuralgia; Neuralgia; Facial Pain | interventions — Pulsed Radiofrequency Treatment; Heart Rate; Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two groups (PRF or PRF + TRF)
Who Masked: Outcomes Assessor
Masking Description: Given the specific nature of the interventions, it may not be possible to blind participants or operators; however, to minimize potential bias, outcome assessors will be blinded to the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Radiofrequency (PRF) (Experimental): Participants in this group will receive pulsed radiofrequency (PRF) treatment targeted to the trigeminal nerve. The procedure will involve a standard PRF protocol.
  Interventions: Procedure: Pulsed Radiofrequency (PRF)
- Pulsed and Thermal Radiofrequency (PRF + TRF) (Active Comparator): Participants in this group will receive a combination of pulsed radiofrequency (PRF) and thermal radiofrequency (TRF). The TRF procedure will involve creating a thermal lesion at a target temperature in addition to the standard PRF treatment protocol.
  Interventions: Procedure: Pulsed and Thermal Radiofrequency (PRF + TRF)

INTERVENTIONS:
Procedure: Pulsed Radiofrequency (PRF) — Participants will receive pulsed radiofrequency (PRF) treatment targeting the trigeminal nerve to manage pain associated with trigeminal neuralgia. This non-ablative technique uses electrical pulses to modulate nerve function, aiming to provide pain relief without creating a thermal lesion.
  Arms: Pulsed Radiofrequency (PRF)
Procedure: Pulsed and Thermal Radiofrequency (PRF + TRF) — Participants will receive a combination of pulsed radiofrequency (PRF) and thermal radiofrequency (TRF) treatments targeting the trigeminal nerve. This approach combines the non-ablative effects of PRF with the thermal lesioning of TRF to provide long-term pain relief for trigeminal neuralgia.
  Arms: Pulsed and Thermal Radiofrequency (PRF + TRF)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of Pulsed Radiofrequency (PRF) with Pulsed and Thermal Radiofrequency (PRF + TRF) in treating Trigeminal Neuralgia (TN) in adults.

The main questions it aims to answer are:

* Does PRF or PRF + TRF provide better pain relief for patients with trigeminal neuralgia?
* What is the safety profile and complication rate of PRF versus PRF + TRF?

Researchers will compare the effects of PRF and PRF + TRF to see if thermal lesioning in addition to pulsed RF provides superior long-term pain relief and reduces the need for analgesic medication.

Participants will:

* Undergo either PRF or PRF + TRF treatment targeting the trigeminal nerve.
* Be assessed for pain relief, functional status, and adverse events over a 3-month follow-up period.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to evaluate the efficacy and safety of Pulsed Radiofrequency (PRF) versus Pulsed and Thermal Radiofrequency (PRF + TRF) for treating Trigeminal Neuralgia (TN). Trigeminal neuralgia is a debilitating chronic pain condition that affects the trigeminal nerve, causing intense facial pain.

The study will enroll participants with TN, randomized into two groups:

* Group 1 (PRF): Patients will receive pulsed radiofrequency treatment with parameters set to standard levels for pain relief.
* Group 2 (PRF + TRF): Patients will receive pulsed radiofrequency combined with thermal lesioning (60-70°C) to target the trigeminal nerve.

Both procedures will be performed under aseptic conditions with appropriate monitoring and anesthesia. The primary outcome will be pain reduction measured using the Numeric Rating Scale (NRS) and Visual Analog Scale (VAS) over a 12-week period. Secondary outcomes include changes in medication consumption assessed by the Medication Quantification Scale III (MQS III) and the recording of procedure-related adverse events.

Participants will undergo follow-up assessments at Week 1, Week 4, and Week 12 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years.
* Diagnosis of classical trigeminal neuralgia, as per the International Classification of Headache Disorders criteria
* Patients experiencing unilateral, episodic facial pain for at least six months with a Numeric Rating Scale (NRS) score greater than 6, despite medical treatment.
* Able to provide informed consent.
* Agree to follow the study procedures and attend follow-up visits.

Exclusion Criteria:

* Patients with secondary trigeminal neuralgia (e.g., due to tumors, multiple sclerosis).
* Previous surgery or radiofrequency treatment for trigeminal neuralgia.
* Pregnant or breastfeeding women.
* Known allergies to anesthetics or other agents used in the procedure.
* Significant psychiatric disorders that may interfere with pain assessment or study participation.
* Coagulopathy or use of anticoagulants that contraindicate the procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Pain Relief - Numeric Rating Scale (NRS) | Baseline, 1 week, 4 weeks, and 12 weeks post-procedure
  The primary outcome measure will be the level of pain relief, assessed using the Numeric Rating Scale (NRS), a scale from 0 to 10, where 0 represents "no pain" and 10 represents "worst possible pain." Pain levels will be recorded at baseline (pre-procedure), and at 1 week, 4 weeks, and 12 weeks post-procedure.
Pain Relief - Visual Analog Scale (VAS) | Baseline, 1 week, 4 weeks, and 12 weeks post-procedure
  Additionally, pain relief will be assessed using the Visual Analog Scale (VAS), a continuous scale ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." Pain levels will be recorded at baseline, 1 week, 4 weeks, and 12 weeks post-procedure.

SECONDARY OUTCOMES:
Medication Consumption | 12 weeks post-procedure
  Changes in medication consumption will be assessed using the Medication Quantification Scale III (MQS III) at 12 weeks post-procedure. This measure evaluates the impact of the interventions on the need for medications to manage trigeminal neuralgia.
Procedure-Related Adverse Events | Immediately post-procedure, 1 week, 4 weeks, and 12 weeks post-procedure
  Adverse events related to the interventions will be systematically recorded to evaluate the safety profile. Adverse events will be monitored and recorded immediately post-procedure and at follow-up visits at 1 week, 4 weeks, and 12 weeks post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Bessar, MD, PhD, Principal Investigator — Assistant Professor of Diagnostic and Interventional Radiology, Zagazig Uni.
Locations (1):
- Zagazig University, Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) with other researchers. This decision is based on considerations related to patient confidentiality, data privacy concerns, and the absence of a current infrastructure for secure data sharing. The primary results of the study will be published in peer-reviewed journals and presented at scientific conferences, ensuring that the findings are accessible to the broader research community.